CLINICAL TRIAL: NCT06633835
Title: Impact of Reactogenicity of the 2024-2025 COVID-19 Vaccines on Health Care Workers and First Responders in the United States
Acronym: SHIELD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019nCoV-415
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Vaccine-Preventable Diseases; SARS CoV 2 Infection
Keywords: COVID-19
MeSH Terms: conditions — COVID-19; Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective interventional study of health care workers (HCW) and first responders (FR) receiving an updated 2024-25 COVID-19 vaccination at the University of Utah (UT). Participants can choose which COVID-19 vaccine type they would like to receive from the study team.
Masking Description: Active comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2024-25 updated Novavax COVID-19 (Active Comparator): Participants will receive a single dose (0.5 ml) of study vaccine Novavax COVID-19 vaccine, 2024-2025 formula (JN.1 containing) in the deltoid muscle of the arm.
  Interventions: Biological: protein subunit: Novavax COVID-19 vaccine
- Pfizer mRNA COVID-19 (Active Comparator): Participants will receive a single dose (0.3 ml) of study vaccine Pfizer mRNA COVID-19 vaccine, 2024-2025 formula (KP.2 containing) in the deltoid muscle of the arm.
  Interventions: Biological: Pfizer mRNA COVID-19 vaccine

INTERVENTIONS:
Biological: protein subunit: Novavax COVID-19 vaccine — Participants will receive a single dose (0.5 ml) of study vaccine Novavax COVID-19 vaccine, 2024-2025 formula (JN.1 containing) in the deltoid muscle of the arm.
  Other Names: 2024-25 COVID-19 vaccination
  Arms: 2024-25 updated Novavax COVID-19
Biological: Pfizer mRNA COVID-19 vaccine — Participants will receive a single dose (0.3 ml) of study vaccine Pfizer mRNA COVID-19 vaccine, 2024-2025 formula (KP.2 containing) in the deltoid muscle of the arm.
  Other Names: 2024-2025 formula
  Arms: Pfizer mRNA COVID-19

SUMMARY:
To assess the impact of reactogenicity among health care workers and first responders receiving an updated 2024-25 Novavax COVID-19 vaccine as compared with those receiving an updated 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine

DETAILED DESCRIPTION:
This is a prospective interventional study of health care workers (HCW) and first responders (FR) receiving an updated 2024-25 COVID-19 vaccination at the University of Utah (UT). Participants can choose which COVID-19 vaccine type they would like to receive from the study team. For this study, health care workers and first responders are defined as anyone having direct face-to-face contact, defined as being within 3 feet, or about an arm's length, with patients as part of their full-time or part-time (greater than or equal to 20 hours per week) job responsibilities.

Approximately 660 health care workers and first responders from Salt Lake City, Utah and surrounding areas will be enrolled into the study. This study will only enroll participants who intend to get an updated 2024-25 COVID-19 vaccine during Fall/Winter 2024-25 SARS-CoV-2 virus circulation. Eligible participants will choose their desired vaccine type (protein subunit: Novavax, or mRNA: Pfizer). Study vaccinators will then administer the chosen vaccine. Following vaccination, study participants will receive a post vaccination questionnaire 48-hours after vaccine administration. Self-reported information on systemic and local reactogenicity symptoms, socio-demographics, occupational history, medical history, COVID-19 and flu vaccine history, and impact on daily activities and work will be collected through the post vaccination questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older who have received at least one COVID-19 vaccination in the past 4 years
* Health care workers or first responders who have direct face-to-face contact, defined as being within 3 feet, or about an arm's length, with patients as part of their full-time or part-time (greater than or equal to 20 hours per week) job responsibilities
* Intends to receive a dose of the updated 2024-25 COVID-19 vaccine
* Able to understand and provide informed consent
* Comfortable reading and responding to text messages and emails sent in English or having an interpreter assist them
* Able and willing to comply with all study requirements
* Access to a smartphone, tablet, or computer to complete the consent, screener and study questionnaires

Exclusion Criteria:

* Ongoing participation in other vaccine or investigational product trials within 90 days of study enrollment
* History of self-reported severe allergic reaction to prior COVID-19 vaccine
* Receipt of COVID-19 vaccine within 60 days of enrollment
* Plans to receive additional vaccines within 7 days after the vaccination visit for study enrollment. (Co-administered vaccinations at time or day of COVID-19 vaccination are permissible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with solicited systemic reactogenicity symptoms. | Day 0 to Day 2
  Percentage of participants that experienced any solicited systemic reactogenicity symptoms after receiving a single dose of 2024-25 Novavax COVID-19 vaccine or 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine during the first two days post vaccination.

SECONDARY OUTCOMES:
Percentage of participants with solicited local reactogenicity symptoms. | Day 0 to Day 2
  To determine the difference in the percentage of participants that experienced any solicited local reactogenicity symptoms after receiving a single dose of 2024-25 Novavax COVID-19 vaccine or 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine during first two days post vaccination.
Number of Participants with solicited systemic reactogenicity symptoms | Day 0 to Day 2
  Number of Participants with solicited systemic reactogenicity symptoms experienced by participants after receiving a single dose of 2024-25 Novavax COVID-19 vaccine or 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine during the first two days post vaccination.
Percentage of participants that experienced multiple solicited systemic reactogenicity symptoms. | Day 0 to Day 2
  Percentage of participants that experienced multiple solicited systemic reactogenicity symptoms after receiving a single dose of 2024-25 Novavax COVID-19 vaccine or 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine during the first two days post vaccination.
Percentage of participants who experienced any local and systemic solicited reactogenicity symptoms. | Day 0 to Day 2
  Percentage of participants who experienced any Local and systemic solicited reactogenicity symptoms that were reported as severity of 2 or higher after receiving a single dose of 2024-25 Novavax COVID-19 vaccine or 2024-25 Pfizer-BioNTech mRNA COVID-19 vaccine during the first two days post vaccination.
Number of Participants Reporting Perceived Impact on Daily Activities (Work, Social, and Family Life) | Day 0 to Day 2
  Number of participants experiencing any perceived impact on their work, social life, and family/home responsibilities within the first 2 days post-vaccination, comparing responses between Novavax and Pfizer-BioNTech mRNA vaccine recipients."

CONTACTS AND LOCATIONS:
Overall Officials: Sarang K Yoon, MOH, Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States